CLINICAL TRIAL: NCT04425928
Title: Comparison of Activity-Based Home Program and Cawthorne-Cooksey Exercises in Patients With Chronic Unilateral Peripheral Vestibular Disorders
Brief Title: Activity Treatment on Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilgehan Tekin Dal (Other)
Responsible Party: Sponsor-Investigator, Bilgehan Tekin Dal, Research Assistant, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 5057087198
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- activity group (Active Comparator): Participants received an activity-based home program that was performed for 4 weeks.
  Interventions: Procedure: occupational therapy based activity training programs
- exercise group (Experimental): Participants received an exercise-based home program was performed that was performed for 4 weeks.
  Interventions: Procedure: Physiotherapy based exercise training programs
- control group (No Intervention): No intervention

INTERVENTIONS:
Procedure: occupational therapy based activity training programs — Occupational therapy based activity training programs in which exercises based on physiotherapy are put into the purposeful activities at vestibular rehabilitation.
  Other Names: purposeful activities
  Arms: activity group
Procedure: Physiotherapy based exercise training programs — Cawthorne-cooksey exercises were performed at vestibular rehabilitation
  Other Names: Cawthorne-cooksey exercises
  Arms: exercise group

SUMMARY:
In this study it was aimed to investigate the effects of home treatment program based standard activity on dizziness, balance and daily life activity in patients with dizziness complaint originated from chronic unilateral peripheral vestibular disorder and compare to effects of exercise-based home rehabilitation program.

DETAILED DESCRIPTION:
The aim of this study was to assess the effects of an activity training programme on dizziness, imbalance, and level of independence in daily living activities in patients with chronic dizziness. 75 patients between 18-65 years of age who diagnosed chronic peripheral vestibular disorders and individuals with vestibular rehabilitation indications were included in our study. Patients were randomly divided into 3 groups consist of 25 patients as an activity group, exercise group, and control group. Education was given to each group. İn addition, the activity group was performed a training activities program, the exercise group was performed in the Cawthorne-Cooksey exercises program. Therapy programs were prescribed once daily at home for 4 weeks. After demographic information was obtained from all patients, assessments were performed at the beginning and at the end of the treatment program (4 weeks). Dizziness severity was assessed by the Visual Analog Scale (VAS), activities of daily livings were assessed by Vestibular Disorders Activity Questionnaire (VADL) and balance was assessed by Sensory Organization Testing (SOT).

ELIGIBILITY:
Inclusion Criteria:

* Patients have dizziness complaint longer than 3 months,
* History of at least one dizziness in a month
* Patient has been diagnosed chronic unilateral peripheric vestibular disorder

Exclusion Criteria:

* Patients with diagnosed benign paroxysmal positional vertigo, had Meniere's disease, had history of central nerve system impairments and/or psychiatric disorder, had uncontrolled hypertension and diabetes, had not understanding simple verbal instruction and following ability, not able to stand independent in the standstill position, had visual problems that cannot be treated with lenses or glasses, had movement limitation due to the orthopedic problem, using medication for dizziness.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Change from before and after treatment in the severity of dizziness on Visual Analog scale (VAS). | before and after treatment (4 weeks)
  VAS is a self-reported instrument assessing the severity of diziness.

SECONDARY OUTCOMES:
Change from before and after treatment in the Independent level of activity in the daily life on Vestibular Disorders Activities of Daily Living Scale (VADL). | before and after treatment (4 weeks)
  VADL is a questionnaire assessing the Independent level of activity in daily life.

OTHER OUTCOMES:
Change from before and after treatment in the postural stability on Computerized Dynamic Posturography (CDP). | before and after treatment (4 weeks)
  Computerized dynamic posturography (CDP) testing is a technique used to assess underlying sensory and motor control impairments associated with balance disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Bumin, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tekin Dal B, Bumin G, Aksoy S, Gunaydin RO. Comparison of Activity-Based Home Program and Cawthorne-Cooksey Exercises in Patients With Chronic Unilateral Peripheral Vestibular Disorders. Arch Phys Med Rehabil. 2021 Jul;102(7):1300-1307. doi: 10.1016/j.apmr.2020.12.022. Epub 2021 Jan 30. PMID 33529612